CLINICAL TRIAL: NCT04136860
Title: Study on the Long-term Outcomes of High-level Cerebral Arteriovenous Malformation
Brief Title: Long-term Outcomes After Different Management Strategies for High-level Cerebral Arteriovenous Malformation
Acronym: OHAVM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, yuanli Zhao, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: KY 2019-09-15
Record Dates: First submitted 2019-09-15; First posted 2019-10-23 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Arteriovenous Malformation of Brain
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Conservative management: Patients refused to accept any interventional treatment or patients were not suitable for any interventional treatment.
- Microsurgical resection: All microsurgical procedures were performed with intraoperative neuronavigation, ultrasonography, indocyanine fluorescence angiography (ICG), continuous monitoring of electroencephalogram and somatosensory evoked potential.
- Embolization: Embolization or radiosurgery was recommended as a priority for lesions located in deep functional locations such as brainstem and basal ganglia. Multi-stage embolization and target embolization were widely used within the embolization. Onyx was the main embolization material.
- Embolization+Radiosurgery: Embolization or radiosurgery was recommended as a priority for lesions located in deep functional locations such as brainstem and basal ganglia. Radiosurgery management was recommended for the residual lesions about 3 months after the embolization if necessary.
- Single-stage hybrid surgery: Hybrid surgery is a new surgical strategy defined as single-stage combined microsurgical resection and embolization in which embolization is performed firstly on the deep feeding artery, aneurysm, AVF, and meningeal arteries involved in blood supply of the nidus, and then, the microsurgical resection was performed immediately. Intraoperative angiography was performed repeatedly before the skull was closed, confirming complete occlusion of the malformation.

SUMMARY:
Arteriovenous malformations (AVMs) are complex and rare cerebral vascular dysplasia. The main purpose of treatment is to avoid the neurological impairment caused by hemorrhagic stroke. The Spetzler-Martin (SM) grading system is widely used to estimate the risk of postoperative complication based on maximum AVM nidus diameter, pattern of venous drainage, and eloquence of location. Generally, grade I and II are amenable to surgical resection alone. Grade III is typically treated via a multimodal approach, including microsurgical resection, embolization, and radiosurgery (SRS). Grade IV and V are generally observed unless ruptured. However, some previous studies indicated that despite the high rate of poor outcomes for high-level unruptured AVMs, the mortality for high-level unruptured AVMs are likely lower than untreated patients. With the development of new embolic materials and new intervention strategies, patients with high-level AVMs may have more opportunities to underwent more aggressive interventions. The OHAVM study aims to clarify the clinical outcomes for patients with SM grade IV and V AVMs after different management strategies.

DETAILED DESCRIPTION:
Follow-up: In our neurosurgical center, follow-up was conducted for all patients at the first 3-6 months and annually after discharge by clinical visit and telephone interview.

Study overview: The population in the OHAVM study will be divided into two parts. Clinical and imaging data of high-level AVM patients from 2012/04 to 2019/09 were retrospectively collected. And the high-level AVM patients from 2019/09 to 2019/12 were prospectively collected. The intervention strategies in our institution for high-level AVMs are of four categories: microsurgical resection, embolization, embolization+radiosurgery, and single-stage hybrid surgery (embolization-resection). Each participants will be followed at least for 5 year since enrollment. Finally, we will clarify the clinical outcomes and prognostic predictors for patients with SM grade IV and V AVMs after different management strategies.

Sample size: About 1000 patients will be enrolled in this study, and half of them were unruptured. The population distribution of different management strategies is expected as follows: conservative:100 cases, microsurgical resection: 300 cases, embolization:250 cases, embolization+radiosurgery: 250 cases, single-stage hybrid surgery: 100 cases.

Study endpoints: The neurological function prognosis, occlusion rate and complications were evaluated at 2 weeks, 1 year, 3 years, 5 years after the treatment and the last follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of AVM was confirmed with digital subtraction angiography (DSA) and/or magnetic resonance imaging(MRI).
2. The SM grade was IV and V.

Exclusion Criteria:

1. Patients with multiple AVMs.
2. Patients with hereditary hemorrhagic telangiectasia (HHT).
3. Patients with missing clinical and imaging data.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Spetzler-Martin (SM) grade IV and V brain arteriovenous malformation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-04-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale score at 2 weeks after the operation | 2 weeks after operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
modified Ranking Scale score at 1 year after the operation | 1 year after operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
modified Ranking Scale score at 3 years after the operation | 3 years after operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
modified Ranking Scale score at 5 years after the operation | 5 years after the operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
modified Ranking Scale score at the last follow-up | up to 10 years after the operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
Long-term hemorrhagic rate | Conservative group: from the diagnosis to the last follow-up (up to 10 years); Intervention group: from 2 weeks after the operation to the last follow-up (up to 10 years)
  For conservative group, the observation period was from the diagnosis to the last follow-up. For the intervention group, to rule out the influence of transient unstable blood flow in the perioperative period, the observation period was defined as from 2 weeks after the operation to the last follow-up.

SECONDARY OUTCOMES:
Obliteration rate | At least 3 years, up to 10 years
  Confirmed by postoperative DSA or MRI/MRA

OTHER OUTCOMES:
Incidence of postoperative epilepsy | 2 weeks and 1 years after the operation and the last follow-up (up to 10 years)
  It can only be diagnosed as postoperative epilepsy with the evidence of typical convulsions and other systemic seizures or EEG evidence.
Incidence of perioperative hemorrhage | 2 weeks after the operation
  Bleeding within two weeks after the operation may be related to the redistribution of cerebral blood flow. The diagnosis of perioperative hemorrhage requires CT confirmation.
Incidence of perioperative infarction | 2 weeks after the operation
  Perioperative infarction within two weeks after the operation may be related to the redistribution of cerebral blood flow. The diagnosis of perioperative infarction requires CT confirmation or MRI confirmation.
Incidence of endovascular embolization injury | 2 weeks after the operation
  Endovascular embolization injuries include arterial dissection, catheter failure, etc.
Incidence of radiation necrosis | Half a year and 1 years after the operation and the last follow-up (up to 10 years)
  Radiation necrosis usually starts to appear within half a year after gamma knife operation. MRI evidence is needed to diagnose radiation necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Capital medical university affiliated Beijing Tiantan hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Chen Y, Li R, Ma L, Meng X, Yan D, Wang H, Ye X, Jin H, Li Y, Gao D, Sun S, Liu A, Wang S, Chen X, Zhao Y. Long-term outcomes of brainstem arteriovenous malformations after different management modalities: a single-centre experience. Stroke Vasc Neurol. 2021 Mar;6(1):65-73. doi: 10.1136/svn-2020-000407. Epub 2020 Sep 14. PMID 32928999
- [Result] Chen Y, Li R, Ma L, Zhao Y, Yu T, Wang H, Ye X, Wang R, Chen X, Zhao Y. Single-Stage Combined Embolization and Resection for Spetzler-Martin Grade III/IV/V Arteriovenous Malformations: A Single-Center Experience and Literature Review. Front Neurol. 2020 Oct 29;11:570198. doi: 10.3389/fneur.2020.570198. eCollection 2020. PMID 33193013
- [Derived] Chen Y, Yan D, Li Z, Ma L, Zhao Y, Wang H, Ye X, Meng X, Jin H, Li Y, Gao D, Sun S, Liu A, Wang S, Chen X, Zhao Y. Long-Term Outcomes of Elderly Brain Arteriovenous Malformations After Different Management Modalities: A Multicenter Retrospective Study. Front Aging Neurosci. 2021 Feb 18;13:609588. doi: 10.3389/fnagi.2021.609588. eCollection 2021. PMID 33679374